CLINICAL TRIAL: NCT07162194
Title: PRIMER (Prostate MRI With Machine LEarning vs. Radiologist) A Novel MRI-Based Machine Learning Approach vs Radiologist MRI Reading for Targeted Prostate Biopsy: A Non-Inferiority, Within-Person Randomized Controlled Trial for Prostate Cancer Detection
Brief Title: MRI-Based Machine Learning Approach Versus Radiologist MRI Reading for the Detection of Prostate Cancer, The PRIMER Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 4P-25-1; NCI-2025-03027 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4P-25-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2025-08-29; First posted 2025-09-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (7):
- Cohort 1 Arm I (MRI/TRUS, PIRADS, GL AI, DL AI) (Experimental): Patients undergo MRI/TRUS followed by a targeted prostate biopsy using PIRADS on study. Patients then undergo a 2nd MRI/TRUS followed by a targeted prostate biopsy based on GL AI predictions. Patients then undergo a 3rd MRI/TRUS followed by a targeted biopsy based on DL AI predictions. Finally, patients undergo up to 12 additional prostate biopsies per SOC.
  Interventions: Procedure: Targeted Prostate Biopsy; Diagnostic Test: Prostate Imaging Reporting & Data System; Diagnostic Test: Deep Learning Artificial Intelligence; Diagnostic Test: Green Learning Artificial Intelligence; Procedure: Radical Prostatectomy
- Cohort 1 Arm II (MRI/TRUS, PIRADS, DL AI, GL AI) (Experimental): Patients undergo MRI/TRUS followed by a targeted prostate biopsy using PIRADS. Patients then undergo a 2nd MRI/TRUS followed by a targeted prostate biopsy based on DL AI predictions. Patients then undergo a 3rd MRI/TRUS followed by a targeted biopsy based on GL AI predictions. Patients undergo up to 12 additional prostate biopsies per SOC. Based on biopsy results, patients will either come off study or undergo radical prostatectomy without hormonal therapy within 180 days from baseline MRI.
  Interventions: Procedure: Targeted Prostate Biopsy; Diagnostic Test: Prostate Imaging Reporting & Data System; Diagnostic Test: Deep Learning Artificial Intelligence; Diagnostic Test: Green Learning Artificial Intelligence; Procedure: Radical Prostatectomy
- Cohort 1 Arm III (MRI/TRUS, GL AI, PIRADS, DL AI) (Experimental): Patients undergo MRI/TRUS followed by a targeted prostate biopsy using GL AI predictions. Patients then undergo a 2nd MRI/TRUS followed by a targeted prostate biopsy using PIRADS. Patients then undergo a 3rd MRI/TRUS followed by a targeted biopsy based on DL AI predictions. Patients undergo up to 12 additional prostate biopsies per SOC. Based on biopsy results, patients will either come off study or undergo radical prostatectomy without hormonal therapy within 180 days from baseline MRI.
  Interventions: Procedure: Targeted Prostate Biopsy; Diagnostic Test: Prostate Imaging Reporting & Data System; Diagnostic Test: Deep Learning Artificial Intelligence; Diagnostic Test: Green Learning Artificial Intelligence; Procedure: Radical Prostatectomy
- Cohort 1 Arm IV (MRI/TRUS, GL AI, DL AI, PIRADS) (Experimental): Patients undergo MRI/TRUS followed by a targeted prostate biopsy using GL AI predictions. Patients then undergo a 2nd MRI/TRUS followed by a targeted prostate biopsy based on DL AI predictions. Patients then undergo a 3rd MRI/TRUS followed by a targeted biopsy using PIRADS. Finally, patients undergo up to 12 additional prostate biopsies per SOC. Patients may also undergo DRE on study.
  Interventions: Procedure: Targeted Prostate Biopsy; Diagnostic Test: Prostate Imaging Reporting & Data System; Diagnostic Test: Deep Learning Artificial Intelligence; Diagnostic Test: Green Learning Artificial Intelligence; Procedure: Radical Prostatectomy
- Cohort 1 Arm V (MRI/TRUS, DL AI, PIRADS, GL AI) (Experimental): Patients undergo MRI/TRUS followed by a targeted prostate biopsy using DL AI predictions. Patients then undergo a 2nd MRI/TRUS followed by a targeted prostate biopsy using PIRADS. Patients then undergo a 3rd MRI/TRUS followed by a targeted biopsy based on GL AI predictions. Patients undergo up to 12 additional prostate biopsies per SOC. Based on biopsy results, patients will either come off study or undergo radical prostatectomy without hormonal therapy within 180 days from baseline MRI.
  Interventions: Procedure: Targeted Prostate Biopsy; Diagnostic Test: Prostate Imaging Reporting & Data System; Diagnostic Test: Deep Learning Artificial Intelligence; Diagnostic Test: Green Learning Artificial Intelligence; Procedure: Radical Prostatectomy
- Cohort 1 Arm VI (MRI/TRUS, DL AI, GL AI, PIRADS) (Experimental): Patients undergo MRI/TRUS followed by a targeted prostate biopsy using DL AI predictions. Patients then undergo a 2nd MRI/TRUS followed by a targeted prostate biopsy based on GL AI predictions. Patients then undergo a 3rd MRI/TRUS followed by a targeted biopsy using PIRADS. Patients undergo up to 12 additional prostate biopsies per SOC. Based on biopsy results, patients will either come off study or undergo radical prostatectomy without hormonal therapy within 180 days from baseline MRI.
  Interventions: Procedure: Targeted Prostate Biopsy; Diagnostic Test: Prostate Imaging Reporting & Data System; Diagnostic Test: Deep Learning Artificial Intelligence; Diagnostic Test: Green Learning Artificial Intelligence; Procedure: Radical Prostatectomy
- Cohort 2 (Radical Prostatectomy Cohort) (Experimental): Patients undergo MRI/TRUS then a radical prostatectomy (RP), which are performed per standard of care at our institution. PIRADS, GL AI, and DL AI will be used to interpret the MRI/TRUS results prior to RP.
  Interventions: Diagnostic Test: Prostate Imaging Reporting & Data System; Diagnostic Test: Deep Learning Artificial Intelligence; Diagnostic Test: Green Learning Artificial Intelligence; Procedure: Radical Prostatectomy

INTERVENTIONS:
Procedure: Targeted Prostate Biopsy — Undergo targeted prostate biopsy
  Other Names: TB; Prostate Biopsy; PBx
  Arms: Cohort 1 Arm I (MRI/TRUS, PIRADS, GL AI, DL AI); Cohort 1 Arm II (MRI/TRUS, PIRADS, DL AI, GL AI); Cohort 1 Arm III (MRI/TRUS, GL AI, PIRADS, DL AI); Cohort 1 Arm IV (MRI/TRUS, GL AI, DL AI, PIRADS); Cohort 1 Arm V (MRI/TRUS, DL AI, PIRADS, GL AI); Cohort 1 Arm VI (MRI/TRUS, DL AI, GL AI, PIRADS)
Diagnostic Test: Prostate Imaging Reporting & Data System — PIRADS Assessment
  Other Names: PIRADS
Diagnostic Test: Deep Learning Artificial Intelligence — Deep Learning (DL) AI predictions
  Other Names: DL AI
Diagnostic Test: Green Learning Artificial Intelligence — Green Learning (GL) AI predictions
  Other Names: GL AI
Procedure: Radical Prostatectomy — Undergo RP
  Other Names: RP

SUMMARY:
This clinical trial studies how well a magnetic resonance imaging (MRI)-based machine learning approach (i.e., artificial intelligence [AI]) works as compared to radiologist MRI readings in detecting prostate cancer. One of the current methods used to help diagnose possible prostate cancer is performing a prostate MRI. An MRI uses a magnetic field to take pictures of the body. The MRI images are examined by a radiologist. If a suspicious area is seen in the MRI, the radiologist assigns it a PIRADS score. This stands for Prostate Imaging Reporting and Data System. The PIRADS score is used to report how likely it is that a suspicious area in the prostate is cancer. The AI system has been developed also to be able to analyze prostate MRI images and detect suspicious areas in the prostate that may be cancer. The AI system's ability to diagnose aggressive prostate cancer may be similar to detection performed by experienced radiologists using the standard PIRADS system of analyzing prostate MRI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the non-inferiority of targeted biopsy according to Green Learning (GL) AI over Prostate Imaging Reporting & Data System (PIRADS).

SECONDARY OBJECTIVES:

I. To determine the clinically significant prostate cancer (CSPCa) detection rate on Deep Learning (DL) AI-targeted biopsy.

II. To determine the patient-level diagnostic performance of GL AI, Deep Learning (DL) AI and PIRADS for clinically significant prostate cancer (CSPCa) detection.

III. To assess Targeted biopsy core characteristics. IV. To evaluate the predictors for patient-level CSPCa detection. V. To assess the spatial correlation of CSPCa distribution on radical prostatectomy (RP) specimens and region of interest (ROI) generated by GL AI and PIRADS.

OUTLINE: Patients undergoing prostate biopsy per standard of care (SOC) are assigned to Group 1. Patients who underwent a prostate biopsy followed by a radical prostatectomy within 6 months, as well as patients only undergoing a radical prostatectomy are assigned to Group 2.

GROUP 1: Patients are randomized to 1 of 6 arms.

ARM I: Patients undergo MRI/transrectal ultrasound (TRUS) followed by a targeted prostate biopsy using PIRADS on study. Patients then undergo a 2nd MRI/TRUS followed by a targeted prostate biopsy based on GL AI predictions. Patients then undergo a 3rd MRI/TRUS followed by a targeted biopsy based on DL AI predictions. Finally, patients undergo up to 12 additional prostate biopsies per SOC.

ARM II: Patients undergo MRI/TRUS followed by a targeted prostate biopsy using PIRADS. Patients then undergo a 2nd MRI/TRUS followed by a targeted prostate biopsy based on DL AI predictions. Patients then undergo a 3rd MRI/TRUS followed by a targeted biopsy based on GL AI predictions. Finally, patients undergo up to 12 additional prostate biopsies per SOC.

ARM III: Patients undergo MRI/TRUS followed by a targeted prostate biopsy using GL AI predictions. Patients then undergo a 2nd MRI/TRUS followed by a targeted prostate biopsy using PIRADS. Patients then undergo a 3rd MRI/TRUS followed by a targeted biopsy based on DL AI predictions. Finally, patients undergo up to 12 additional prostate biopsies per SOC.

ARM IV: Patients undergo MRI/TRUS followed by a targeted prostate biopsy using GL AI predictions. Patients then undergo a 2nd MRI/TRUS followed by a targeted prostate biopsy based on DL AI predictions. Patients then undergo a 3rd MRI/TRUS followed by a targeted biopsy using PIRADS. Finally, patients undergo up to 12 additional prostate biopsies per SOC.

ARM V: Patients undergo MRI/TRUS followed by a targeted prostate biopsy using DL AI predictions. Patients then undergo a 2nd MRI/TRUS followed by a targeted prostate biopsy based on GL AI predictions. Patients then undergo a 3rd MRI/TRUS followed by a targeted biopsy using PIRADS. Finally, patients undergo up to 12 additional prostate biopsies per SOC.

ARM VI: Patients undergo MRI/TRUS followed by a targeted prostate biopsy using DL AI predictions. Patients then undergo a 2nd MRI/TRUS followed by a targeted prostate biopsy using PIRADS. Patients then undergo a 3rd MRI/TRUS followed by a targeted biopsy based on GL AI predictions. Finally, patients undergo up to 12 additional prostate biopsies per SOC.

GROUP 2: Patients have their removed prostate evaluated using a special mold on study. Prostate tissue is mapped and compared with the prostate cancer prediction on MRI generated by radiologists and AI reports.

After completion of study intervention, patients are followed up at 10 days and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* PROSTATE BIOPSY COHORT: Patients undergoing transperineal MRI/TRUS fusion prostate biopsy (PBx) as per standard of care
* PROSTATE BIOPSY COHORT: Patients who underwent or are undergoing 3T multiparametric MRI (T2W, diffusion weighted imaging [DWI], apparent diffusion coefficient [ADC], and dynamic contrast-enhanced [DCE]) within 90 days prior to biopsy
* PROSTATE BIOPSY COHORT: Patients who consented to the study
* RADICAL PROSTATECTOMY COHORT: Patients undergoing radical prostatectomy for primary treatment of prostate cancer as per standard of care
* RADICAL PROSTATECTOMY COHORT: Patients who underwent or are undergoing 3T multiparametric MRI (T2W, DWI, ADC, and DCE) within 180 days prior to radical prostatectomy
* RADICAL PROSTATECTOMY COHORT: Patients who consented to the study

Exclusion Criteria:

* PROSTATE BIOPSY COHORT: Patients with a history of prostate cancer
* PROSTATE BIOPSY COHORT: Patients with a history of surgical treatment on benign prostate hyperplasia
* PROSTATE BIOPSY COHORT: Patients undergoing saturation prostate biopsy
* PROSTATE BIOPSY COHORT: Patients under 20 years old
* PROSTATE BIOPSY COHORT: Patients with previous PBx history
* PROSTATE BIOPSY COHORT: MRI which was not interpreted by PIRADS
* PROSTATE BIOPSY COHORT: MRI with significant artifact
* RADICAL PROSTATECTOMY COHORT: Patients who are undergoing neo-adjuvant hormonal therapy in conjunction with radical prostatectomy
* RADICAL PROSTATECTOMY COHORT: Patients with a history of surgical treatment on benign prostate hyperplasia
* RADICAL PROSTATECTOMY COHORT: Patients under 20 years old
* RADICAL PROSTATECTOMY COHORT: Patients without pre-treatment MRI
* RADICAL PROSTATECTOMY COHORT: MRI which was not interpreted by PIRADS
* RADICAL PROSTATECTOMY COHORT: MRI with significant artifact
* RADICAL PROSTATECTOMY COHORT: Patients who are included in the Biopsy cohort

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2028-10-15 (Estimated)

PRIMARY OUTCOMES:
Clinically-significant prostate cancer (CSPCa) detection rate on Green Learning (GL) artificial intelligence (AI)-targeted and Prostate Imaging-Reporting and Data System (PIRADS)-targeted biopsies | Up to 3 months
  Detection rates of PIRADS and GL AI-targeted biopsy will be evaluated per index region of interest (ROI), respectively.
CSPCa detection rate on GL AI-targeted and Deep Learning (DL) AI-targeted biopsies | Up to 3 months
  Detection rates of GL AI and DL AI targeted biopsy will be evaluated per index ROI, respectively.

SECONDARY OUTCOMES:
Patient-level diagnostic performance of GL AI and PIRADS for CSPCa detection | Up to 3 months
  Sensitivity, specificity, accuracy, positive predictive value, and negative predictive value will be compared between PIRADS, GL AI, and DL AI predictions by McNemar test. The performance will be calculated according to the definitions below. Additionally, decision curve analysis will be conducted.
Targeted biopsy core characteristics | Up to 3 months
  Will include prostate cancer subtypes, benign elements, lesion locations, cancer core length (mm), cancer core involvement (%), and Gleason Grade Group. Will be compared between PIRADS, GL AI, and DL AI by Chi-square test or Wilcoxon rank sum test.
Predictors for patient-level CSPCa detection | Up to 3 months
  Independent predictors for patient-level CSPCa detection will be assessed by logistic regression. Predictors include age, race, ethnicity, prostate-specific antigen (PSA), PSA density (PSA/prostate volume measured on magnetic resonance imaging [MRI]), digital rectal examination (DRE) abnormality, PIRADS score, GL AI prediction score, and DL AI prediction score. Classifier will be created using the strong predictors for CSPCa, and its discriminant performance will be assessed by the receiver operating characteristic (ROC) analysis.
Dice score and linear correlation coefficient of CSPCa distribution on radical prostatectomy (RP) specimens and ROI generated by GL AI, DL AI and PIRADS | Up to 3 months
  Distribution of CSPCa on the RP specimen will be annotated on the digitized slides and 3-dimensional reconstructed as ground truth. ROI segmentations according to PIRADS, GL AI prediction heatmap, and DL AI prediction heatmap also will be 3D reconstructed. The spatial concordance between GL-ROI, DL AI-ROI, PIRADS-ROI, and CSPCa distribution on RP specimen will be assessed. The accuracy of the spatial concordance and volume estimation will be analyzed by the Dice score and linear correlation analysis, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Luis Abreu, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States